CLINICAL TRIAL: NCT01098513
Title: Relative Bioavailability Study of Three Different Tablet Formulations of GSK1349572 50 mg and the Dose Proportionality of and Effect of Food on the Selected Formulation in Healthy Male and Female Volunteers (ING113674)
Brief Title: GSK1349572 Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113674
Record Dates: First submitted 2010-03-25; First posted 2010-04-02 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2011-02

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: HIV; healthy; GSK1349572
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will be randomized in a three-way crossover design to receive a single dose of each of three different tablet formulations of GSK1349572 50 mg (2 tablets). Formulation AP, AW and AX.
  Interventions: Drug: GSK1349572 formulation AP; Drug: GSK1349572 formulation AW; Drug: GSK1349572 formulation AX
- Part B (Experimental): A total of 18 subjects who complete Part A will return for Part B. Subjects from Part A will be asked to participate on a first come first served basis until there are 18 subjects, at which time enrolment to Part B will be closed. Part B will be a three way crossover design using either formulation AW or AX depending upon the results from Part A. Subjects will receive a single dose of 50 mg GSK1349572 with either a low fat, moderate fat or high fat meal in each period.
  Interventions: Drug: GSK1349572 formulation AW; Drug: GSK1349572 formulation AX

INTERVENTIONS:
Drug: GSK1349572 formulation AP — GSK1349572 50 mg single dose fasted.
  Arms: Part A
Drug: GSK1349572 formulation AW — GSK1349572 formulation AW 50 mg single dose in Part A and 75 to 200 mg fasted or with moderate or high fat meal in Part B.
Drug: GSK1349572 formulation AX — GSK1349572 formulation AX 50 mg in Part A and 75-200 mg fasted or with a moderate or high fat meal in Part B

SUMMARY:
This is a single-center, randomized, two part, open-label, crossover study in healthy adult subjects. Part A will evaluate the relative bioavailability of two new tablet formulations compared to the current tablet formulation of GSK1349572 at 50 mg administered as single doses each comprising of two 25 mg tablets. Pharmacokinetic samples from Part A will be analyzed and, if at least one of the new formulations meets appropriate criteria and is selected, Part B will be a single-sequence design conducted to evaluate food effect of the selected new tablet formulation at one dose level. A subset of subjects enrolled in Part A will continue in Part B. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-28 days after the last dose of study drug.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equla to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<146.8 pmol/L) is confirmatory] or Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 AUC(0-infinity), AUC(0-t), and Cmax. | 48 hours

SECONDARY OUTCOMES:
Plasma GSK1349572 t½, tlag, tmax, C24, Vdss/F, CL/F, and MRT. | 48 hours
Safety and tolerability parameters, including adverse events, concurrent medication, clinical laboratory screens, ECG, and vital signs assessments. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States